CLINICAL TRIAL: NCT03482869
Title: The Walking Estimated Limitation Stated by History (WELSH): A Visual Tool to Self-report Walking Impairment From a Predominantly Illiterate Diabetic Population.
Brief Title: Evaluation of Self-reported Walking Impairment in Predominantly Illiterate Patients
Acronym: WELSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Polytechnique de Bobo-Dioulasso (Other)
Responsible Party: Principal Investigator, Nafi OUEDRAOGO, Head of department of physiology, Université Polytechnique de Bobo-Dioulasso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Bobo 2018-001
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Diabetes
Keywords: walking impairment; disability; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetic patients (Experimental): Patients referred for the equilibrium or diagnosis of diabetes mellitus will be proposed to participate and estimate their walking ability with the WELSH (Walking estimated limitation stated by History) based solely on images
  Interventions: Diagnostic Test: walking ability

INTERVENTIONS:
Diagnostic Test: walking ability — Included patients will perform a 6 min walk test

SUMMARY:
The purpose of this study is to test the routine feasibility of an image tool adapted from the WELCH questionnaire ( Walking estimated limitation calculated by history) to estimate walking impairment (The WELSH questionnaire: Walking estimated limitation stated by history) in patients investigated for walking impairment. Secondary aims correlation with the maximal walking distance.

DETAILED DESCRIPTION:
The WELSH is self completed by the patients and scored by the physician after self-completion. Patients perform a 6 minutes walking test on a 30m corridor

ELIGIBILITY:
Inclusion Criteria:

* •Signed consent for the data treatment as a database

Exclusion Criteria:

* Rebuttal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-30 (Estimated); Primary Completion 2018-08-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance | 10 minutes
  Maximal measured distance will be the distance walked during a 6 min walk tests

CONTACTS AND LOCATIONS:
Overall Officials: Nafi OUEDRAOGO, Principal Investigator — CHU Souro Sanou
Locations (1):
- CHU Souro Sanou, Bobo-Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: Undecided
Probably available upon request. Undecided yet